CLINICAL TRIAL: NCT06259019
Title: Site of Disease BIOmolecule Capture and Analysis in PATienTs With Established Coronary Disease undERgoing iNtracoronary Assessment
Brief Title: Liquid Biopsy System Intracoronary Blood Sampling and Analysis to Characterise Disease Biomarkers in Patients With Coronary Disease
Acronym: BIOPATTERN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PlaqueTec Ltd (Industry)
Collaborators: Royal Papworth Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 65112021
Record Dates: First submitted 2023-12-12; First posted 2024-02-14 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: Liquid Biopsy System; Intracoronary; Biomarkers; PlaqueTec; BIOPATTERN
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liquid Biopsy System (Other): Main trial arm, all recruited and enrolled patients will undergo intracoronary blood sampling using the Liquid Biospy System Device.
  Interventions: Device: Liquid Biopsy System (LBS)

INTERVENTIONS:
Device: Liquid Biopsy System (LBS) — Coronary artery catheter designed to mix intra-arterial flow and simultaneously extract multiple blood samples from around the site of coronary disease within a vessel of interest.
  Other Names: LBS

SUMMARY:
The aim of this research, proposed and funded by PlaqueTec and co-ordinated by Papworth Trials Unit Collaboration, is to demonstrate the performance of the coronary artery blood sampling device (Liquid Biospy System, LBS) and establish its usefulness to collect a range of disease biomolecules from the coronary artery of interest. Using the data generated from extensive analysis of the blood samples, key biomarker data will be generated that will close a knowledge gap and facilitate the development of tailored treatments for coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

Stage 1 screening inclusion:

1. ≥18 years of age, have capacity and be willing to provide informed consent to participate
2. Clinical evidence of obstructive coronary artery disease and be scheduled for either:

   1. Elective coronary angiography +/- proceed for stable angina OR
   2. Elective PCI for stable angina with known bystander disease not for PCI OR
   3. Angiography +/- proceed for Troponin negative unstable angina

Stage 2 screening inclusion:

Suitable lesion identified meeting angiographic criteria for LBS deployment and Cardiologist comfortable to deploy OCT and LBS on study lesion before carrying out PCI on any other lesion

Exclusion Criteria:

Stage 1 screening exclusion:

1. Myocardial Infarction within 30 days of procedure.
2. Chronic renal failure (eGFR<30ml/min/1.73m2).
3. Contrast allergy.
4. Hypotension, shock or haemodynamic instability.
5. Ventricular arrhythmia.
6. Chronic Heart Failure (NYHA ≥ 3) or LVEF ≤ 30%.
7. Immunocompromised or receiving immunosuppressant therapy.
8. Any active disease that in the opinion of the investigator makes the subject unsuitable for the research procedure or subject life expectancy less than 1 year.
9. Active infection or sepsis (significant CRP elevation and/or requiring antibiotics).
10. Active systemic inflammatory condition.
11. Inability to receive anticoagulants or antiplatelets or uncorrected bleeding disorder or deranged platelet count.
12. Is pregnant.
13. Deemed high clinical risk or unsuitable for the procedure for any reason by the treating clinician.

Stage 2 screening exclusion:

1. Target lesion is in the left main coronary artery.
2. Target lesion requires PCI
3. In same vessel as lesion requiring PCI
4. Unsuitable coronary anatomy (vessel tortuosity [>45 degree bend], moderate/ severe calcification angiographically, ostial disease).
5. Presence of thrombus in the target vessel.
6. Prior PCI or stent in vessel identified for LBS sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Trans-plaque gradients (downstream value divided by upstream value) for LOX-1 and CXCL1 | Single time point (time of intervention)
Liquid Biopsy System (LBS) performance: successful positioning and successful intracoronary sampling | Single time point (time of intervention)
  Success define as confirmed adequate positioning of the device across the identified lesion of interest and collection of sufficient whole blood from each functional port to generate >100µl plasma once processed

SECONDARY OUTCOMES:
Correlations between primary outcome measure proteins and: patient subsets and lesion level data | Single time point (time of intervention)
  Patient level subsets:
  * With and without type 2 diabetes mellitus
  * Prior/no prior history of Myocardial Infarction (MI)
  Lesion level data:
  - Coronary fibroatheroma cap thickness and lipid arc as measured by OCT image analysis

OTHER OUTCOMES:
Incidence of adverse events in subjects in whom the LBS is used | During intervention and subsequent 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Steve Hoole, Principal Investigator — Royal Papworth Hospital NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Heart Institute, Bristol
  - Royal Papworth Hospital, Cambridge
  - Norfolk and Norwich Hospital, Norwich

IPD SHARING:
Plan to Share IPD: No